CLINICAL TRIAL: NCT03797755
Title: Prospective Observational Study of the Prognosis of Patients Having Palliative Radiotherapy
Brief Title: Prognosis of Patient Evaluated for Palliative Radiotherapy
Acronym: PROPER
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tuen Mun Hospital (Other Government)
Responsible Party: Principal Investigator, Shing Fung Lee, Resident Specialist, Tuen Mun Hospital
Other Study IDs: NTWC_Onc_2019
Record Dates: First submitted 2019-01-07; First posted 2019-01-09 (Actual); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Cancer; Radiotherapy
Keywords: survival; cancer; palliative; radiotherapy; prognosis
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Palliative Cancer Patients: Stage IV cancer patients evaluated for palliative radiotherapy.
  Interventions: Radiation: palliative radiotherapy

INTERVENTIONS:
Radiation: palliative radiotherapy — Radiotherapy for palliating symptoms in stage IV cancer patients

SUMMARY:
Many patients with incurable cancer will receive palliative oncological treatment before their death, and radiotherapy (RT) is an important element of this. The aim of palliative RT is to alleviate symptoms and improve quality of life. An accurate and practical survival prediction model for metastatic cancer patient receiving palliative RT can assist the decision making (ranging from best supportive treatment alone for expected short survival, to dose escalation for potential better disease control).

The available survival prediction models (such Survival Prediction Score using Number of Risk Factors by Chow et al and TEACHH model) have been developed in the Western world. We therefore perform a prospective observational study 1) to assess the overall survival of patients evaluated for palliative RT at a tertiary hospital in Hong Kong, and 2) to validate the prognostic score systems in our population.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients with stage IV cancer who are referred for palliative RT in Tuen Mun Hospital, including both inpatients and outpatients.

Exclusion Criteria:

* Patients who have received palliative RT before (i.e. not the first course palliative RT), have non-metastatic disease, are misclassified as palliative patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stage IV cancer patients evaluated for palliative radiotherapy in Tuen Mun Hospital
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 1 year
  Overall Survival in the studied population

SECONDARY OUTCOMES:
Overall Survival in Each Indication of Palliative Radiotherapy | 3, 6, 9, 12 months
  Indications of Palliative Radiotherapy:
  The indication will be as follow:
  spinal cord compression brain metastases tumor bleeding tumoral mass Cancer pain Superior Vena Cava Syndrome/ Airway compression
Overall Survival by Survival Prediction Model (NRF) | 3, 6, 9, 12 months
  Overall Survival by Survival Prediction Score using Number of Risk Factors (NRF)
Overall Survival by Survival Prediction Model (TEACHH) | 3, 6, 9, 12 months
  Overall Survival by Survival Prediction Score using TEACHH Model

CONTACTS AND LOCATIONS:
Overall Officials: Shing Fung Lee, MBBS (HK), FRCR (UK), Principal Investigator — Department of Clinical Oncology, New Territory West Cluster, Hospital Authority, Hong Kong
Locations (1):
- Department of Clinical Oncology, Tuen Mun Hospital, Tuen Mun, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Demographic data, and the information required for the prognostic scores will be extracted (e.g. presence of liver metastasis). Also data on the date of birth and death, sex, primary cancer. Data on the primary site of disease were coded using International Classification of Disease version 9.
  Personal identifier will be deleted to protect patient confidentiality.
Supporting Information: Analytic Code
Time Frame: After publication.

REFERENCES:
- [Background] Chow E, Harth T, Hruby G, Finkelstein J, Wu J, Danjoux C. How accurate are physicians' clinical predictions of survival and the available prognostic tools in estimating survival times in terminally ill cancer patients? A systematic review. Clin Oncol (R Coll Radiol). 2001;13(3):209-18. doi: 10.1053/clon.2001.9256. PMID 11527298
- [Background] Christakis NA, Lamont EB. Extent and determinants of error in doctors' prognoses in terminally ill patients: prospective cohort study. BMJ. 2000 Feb 19;320(7233):469-72. doi: 10.1136/bmj.320.7233.469. PMID 10678857
- [Background] Gripp S, Mjartan S, Boelke E, Willers R. Palliative radiotherapy tailored to life expectancy in end-stage cancer patients: reality or myth? Cancer. 2010 Jul 1;116(13):3251-6. doi: 10.1002/cncr.25112. PMID 20564632
- [Background] Chow E, Abdolell M, Panzarella T, Harris K, Bezjak A, Warde P, Tannock I. Predictive model for survival in patients with advanced cancer. J Clin Oncol. 2008 Dec 20;26(36):5863-9. doi: 10.1200/JCO.2008.17.1363. Epub 2008 Nov 17. PMID 19018082
- [Background] Peppercorn JM, Smith TJ, Helft PR, Debono DJ, Berry SR, Wollins DS, Hayes DM, Von Roenn JH, Schnipper LE; American Society of Clinical Oncology. American society of clinical oncology statement: toward individualized care for patients with advanced cancer. J Clin Oncol. 2011 Feb 20;29(6):755-60. doi: 10.1200/JCO.2010.33.1744. Epub 2011 Jan 24. PMID 21263086
- [Background] Chow E, James JL, Hartsell W, Scarantino CW, Ivker R, Roach M III, Suh JH, Demas W, Konski A, Bruner DW. Validation of a Predictive Model for Survival in Patients With Advanced Cancer: Secondary Analysis of RTOG 9714. World J Oncol. 2011 Aug;2(4):181-190. doi: 10.4021/wjon325w. Epub 2011 Aug 24. PMID 29147245
- [Background] Krishnan MS, Epstein-Peterson Z, Chen YH, Tseng YD, Wright AA, Temel JS, Catalano P, Balboni TA. Predicting life expectancy in patients with metastatic cancer receiving palliative radiotherapy: the TEACHH model. Cancer. 2014 Jan 1;120(1):134-41. doi: 10.1002/cncr.28408. Epub 2013 Oct 2. PMID 24122413